CLINICAL TRIAL: NCT04642066
Title: Effect of Repeatedly Applied Cold Water Immersion on Subclinical Atherosclerosis, Inflammation, Fat Accumulation and Lipid Profile Parameters of Volunteers
Brief Title: Cold Water Immersion and Atherosclerosis, Inflammation, Fat Accumulation and Lipid Profile Parameters
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not obtained
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Martin Janičko, Assistant Professor, Pavol Jozef Safarik University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LF UPJS
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Risk Factor; Metabolic Complication; Endocrine; Complications; Immune System Diseases
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Healthy volunteers were followed during the 5-month CWI exposition under standard conditions (three times per week 7-10 min). Neoprene equipment was not allowed; volunteers with followed weight or muscle mass changes over 5% were excluded
  Interventions: Other: Cold water immersion
- Sham control (Sham Comparator): Control without CWI exposition
  Interventions: Other: No cold water immersion

INTERVENTIONS:
Other: Cold water immersion — Full body CWI in open standing, except the head (same location, timing), frequency three times a week in the duration of 7-10 minutes. Swimming was permitted. Volunteers must not use neoprene aids (gloves, shoes), caps were allowed. Volunteers should be in the final phase submerged in water, above which there should only be the head and neck. The upper limbs were below the water surface. Non-neoprene footwear was permitted. Volunteers entered the water continuously without stopping. The time of stay in water was calculated from the first contact of the foot with water. On average, the whole body needed to be immersed in water within 30 seconds.
  Arms: Active Group
Other: No cold water immersion — People without cold water immersion
  Arms: Sham control

SUMMARY:
The impact of the environment on human health is considerable. An important factor is the effect of temperature on the human body, where either the effects of short-term exposure to extreme temperatures (cryotherapy, sauna, etc.) or the long-term environmental impact are monitored.

The study was focused on research of the long-term effect of repeated CWI on atherogenesis, lipid parameters and fat distribution.

DETAILED DESCRIPTION:
This study was designed as a cohort observational studyfollowing the group of volunteers practicing CWI. Totally forty volunteers agreed to participate in the study by signing the informed consent, approved by the local ethics committee of UPJŠ Košice. Volunteers were examined in Cardiology and General Medicine outpatient clinics of Faculty of medicine, UPJŠ Košice (1st Department of Internal Medicine; outpatient clinics of Medicomp Košice Ltd.). They underwent the anamnesis and examination with a focus in the first step on matching the inclusion criteria: SCORE for the assessment of the cardiovascular risk as low (≤1%), patients without the suspected diagnosis of the familialhypercholesterolemia, respectively with TC level above 8 mmol/L, respectively TG concentrations above 2.3 mmol/L, male gender, age between 21 and 60, signed informed consent to participate in the study.

Patients with one or more exclusion criteria were not included: volunteers with lipid-lowering therapy or those that received hypolipidemics in the period shorter than 3 months before the study, values of blood lipids outside the inclusion criteria, glucose intolerance and DM,presence of advanced cardiovascular (plague or coronary artery disease, TIA, stroke, etc.) or chronic inflammatory diseases, infection or diseases possible affecting measured parameters and significant lifestyle changes in the last period of 6 months before the CWI.

After the initial examination, 35 volunteers fulfilled the criteria. Volunteers of the study underwent controlled, repeated CWI (5 months 15/11/18 - 15/03/19)based on a following pre-prepared protocol in the cooperation of our physicians and the sport club: Full body CWI in open standing, except the head (same location, timing), frequency three times a weekin the duration of 7-10 minutes. Swimming was permitted. Volunteers must not use neoprene aids (gloves, shoes), caps were allowed. Volunteers should be in the final phase submerged in water, above which there should only be the head and neck. The upper limbs were below the water surface. Non-neoprene footwear was permitted. Volunteers entered the water continuously without stopping. The time of stay in water was calculated from the first contact of the foot with water. On average, the whole body needed to be immersed in water within 30 seconds. The entire study was performed in the nearby lake, where all participants in the active arm were exposed to the same weather and water conditions, which were monitored. Volunteers who did not follow the protocol in more than 15% of the episodes, respectively, with weight, fat or muscle mass changes over 5%, with significant dietary changes were excluded from the study. Equivalent sham control group (N=30) was included fulfilling the inclusion criteria, without the CWI.

ELIGIBILITY:
Inclusion Criteria:

without cardiovascular and metabolic disease cold water immersion

Exclusion Criteria:

cancer inflammatory diseases cardovascular diseases tuberculosis renal and hepatic insufficiency pregnancy cardiovascular diseases obesity metabolic syndrome lymphoproliferative disorders liver transplantation in the past suspected. chronic infection in risk locations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 6 months
  BMI kg/m2
Change in total cholesterol from baseline | 6 months
  percentual change in total cholesterol (mmoL/L)
Concentrations of PCSK9, hsCRP and other inflammation markers | 6 months
  mmol/l
cIMT | 6 months
  mm
PWV | 6 months
  m/s
Beta | 6 months
AU | 6 months
SF | 6 months
  mm
VF | 6 months
  mm
Fatty acid profile | 6 months
  mol/l

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Tóth, MUDr., PhD, Principal Investigator — Pavol Joef Safárik University, Faculty of Medicine
Locations (1):
- 1st Department of Internal medicine, L. Pasteur University Hospital in Košice, Košice, Slovakia